CLINICAL TRIAL: NCT02463318
Title: The Effect of Melatonin on Gene Expression and Activity of the Sirt1 and Its Target Genes Catalase and MnSOD in Multiple Sclerosis Patients and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 91-01-30-17019
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2015-06

CONDITIONS: Multiple Sclerosis; Oxidative Stress
Keywords: Multiple sclerosis; SIRT1; MnSOD; Catalase; Oxidative stress; Antioxidant enzyme
MeSH Terms: conditions — Multiple Sclerosis | interventions — Melatonin; Hydrogen Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple slerosis (Experimental): Melatonin,,one millimolar,one micromolar,one nanomolar, 12 hr treatment.
  Interventions: Drug: Melatonin
- Healthy subjects (Experimental): Melatonin,one millimolar,one micromolar,one nanomolar, 12 hr treatment. hydrogen peroxide, 250 micromollar,2 hr treatment
  Interventions: Drug: Melatonin; Other: Hydrogen peroxide

INTERVENTIONS:
Drug: Melatonin — Melatonin is used for healthy subjects and multiple sclerosis patients
  Other Names: N-acetyl-5-methoxy tryptamine
Other: Hydrogen peroxide — Hydrogen peroxide is only used for healthy subjects
  Arms: Healthy subjects

SUMMARY:
The purpose of this study is to investigate the gene expression and activity of SIRT1, and forkhead box O3 pathway by means of investigating target genes MnSOD and catalase in multiple sclerosis and healthy subjects. Also, we investigate the effect of melatonin on interaction between SIRT1 activity and target genes MnSOD and catalase in multiple sclerosis and healthy subject .Additionally, we evaluate effect the probable effect of melatonin treatment on gene expression and activity of above-mentioned genes in peripheral blood mononuclear cells of healthy subjects-treated with H2O2.

ELIGIBILITY:
Inclusion Criteria:

patients with relapsing-remitting multiple sclerosis. The diagnosis of MS was based on the McDonald criteria . All patients were newly diagnosed cases with an Expanded Disability Status Scale (EDSS) score ≤ 6 and had never received immunomodulatory and immunosuppressive drugs.

-

Exclusion Criteria:

* The exclusion criteria were as follows: 1) treated with antioxidant supplements, anti-inflammatory drugs, and vitamins in the previous 6 months; 2) had a history of acute or chronic infection, malignancy, diabetes (type I and II), and any clinically significant systemic disease; 3) was currently pregnant or lactating; 4) was currently smoking; 5) used contraceptive medication during the previous 6 months.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Relative gene expression by real-time PCR (polymerase chain reaction) | Change from baseline after 12-hour treatment with melatonin and 2 -hours treatment with H2O2

SECONDARY OUTCOMES:
MnSOD enzyme activity assay | Change from baseline after 12-hour treatment with melatonin and 2 -hours treatment with H2O2
Catalse enzyme activity assay | Change from baseline after 12-hour treatment with melatonin and 2 -hours treatment with H2O2
SIRT1 enzyme activity assay | Change from baseline after 12-hour treatment with melatonin and 2 -hours treatment with H2O2

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Sahraian, Neurologist, Study Director — Tehran University of Medical Sciences; Solaleh Emamgholipour, PhD Student, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Solaleh Emamgholipour, Tehran, Iran